CLINICAL TRIAL: NCT01683500
Title: Calcinosis Cutis: Therapeutic Effects of Extracorporeal Shock Wave Therapy (ESWT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCESWT01
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Calcinosis Cutis in Connective Tissue Disease
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- shock wave therapy (Experimental): intervention: shock wave therapy with Modulith SLK (Storz)
  Interventions: Device: shock wave therapy with Modulith SLK (Storz)

INTERVENTIONS:
Device: shock wave therapy with Modulith SLK (Storz) — Three sessions with shock wave therapy, interval of one week.

SUMMARY:
Patients with calcinosis cutis due to connective tissue disease get a shock wave therapy. The shock wave therapy will be done in 3 sessions with one week interval. The outcome parameters are: change in pain, size of the calcinosis, of possible ulcers and intake of painkillers.

* Trial with medical device

DETAILED DESCRIPTION:
Patients with calcinosis cutis due to connective tissue disease get a shock wave therapy (medical device). The shock wave therapy will be done in 3 sessions with one week interval. The outcome parameters are: change in pain (questionnaire), size of the calcinosis (ultrasound and CT), new ulcers and intake of painkillers.

ELIGIBILITY:
Inclusion criteria:

* Age of 18
* Calcinosis cutis due to connective tissue disease
* information about ESWT given
* Patient understands the study and signs the informed consent

Exclusion criteria:

* No ESWT done
* cuagulopathy
* sepsis
* pregnancy
* pace maker
* severe disease in the opinion of the investigator
* cardiac risk with NYHA III-IV
* Ehlers-Danlos-Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
change in pain | after 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Blumhardt, MD, Principal Investigator — University Hospital Zurich, Division of Rheumatology
Locations (1):
- University Hospital Zurich, Division of Rheumatology, Zurich, Canton of Zurich, Switzerland